CLINICAL TRIAL: NCT04037150
Title: Circulating DNA in Non-small Cell Lung Cancer Patients: Relation to Tumor Burden, Disease Prognosis and Risk for Cancer Recurrence, With Emphasis on Tumor Heterogeneity and Treatment Response
Brief Title: Circulating DNA in Surgically Treated NSCLC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Institute for Molecular Medicine (Other)
Responsible Party: Principal Investigator, Ilkka Ilonen, Principal Investigator, Helsinki University Central Hospital
Other Study IDs: Y2019SK007
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; cfDNA
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Circulating tumor DNA and tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Circulating tumor DNA — Circulating tumor DNA

SUMMARY:
* The investigators will prospectively recruit 100 NSCLC patients. The cfDNA samples will be gathered before the surgery and postoperatively 4-6 weeks after surgery and at 6 and 12 months follow-up visits.
* This study aims to investigate the role of ctDNA in NSCLC patients treated with curative intent surgery.
* Preoperative ctDNA will be compared to primary tumor DNA to investigate the concordance of mutations and gained mutations from possible primary tumor cancer stem cell.
* Preoperative ctDNA findings will be tested for associations with baseline characteristics as well as clinically important factors such as TNM stage, histopathological findings, and tumor volume.
* The investigators aim to identify molecular residual disease (MRD) using multiple ctDNA samples after the surgery and search the associations with clinical recurrence and survival, with possible correlation to palliative chemotherapy response
* Using multiple ctDNA samples, the investigators will gather information about tumor heterogeneity, diversity of disease genotypes, and dynamic changes in ctDNA.
* If additional data from palliative immunotherapy (PD-L1 inhibitors) is available, the effect of this will be evaluated in the study.

DETAILED DESCRIPTION:
Plasma liquid biopsy is rapidly emerging non-invasive diagnostic tool that could be used as a surrogate for tumor biopsy or disease activity. Circulating cell-free DNA (cfDNA) is short fragment double stranded DNA that is present in blood. Ultrasensitive mutation specific techniques based on polymerase-chain-reaction (PCR) analysis are required to detect mutations and alterations in circulating tumor cells. Early studies based on a small number of patients indicate that ctDNA analyses could be used for molecular testing, cancer detection, surrogate for tumor burden or activity, and treatment monitoring in solid tumors.

In the current study the role of ctDNA from plasma in surgically treated early stage NSCLC patients will be investigated. The investigators aim to collect a prospective cohort of a hundred patients with preoperative and follow-up samples as well as diagnostic tissue specimen. The investigators hypothesize that longitudinal ctDNA-samples could be used as prognostic marker for recurrence and survival. Finding postsurgical positive ctDNA could aid us to identify patients who would benefit from adjuvant chemotherapy before clinical recurrence.

Study design and ethical considerations

This is a prospective, non-interventional, single arm study that will be conducted in collaboration with Helsinki Biobank. It is estimated that cohort of 100 patients will provide with ample sample size, as 30-40% will develop a recurrence during the 5 year follow up. A preliminary agreement with Helsinki Biobank about the sample collection and storage has been made. There will be no additional study appointments as all the control visits and study samples are scheduled according to normal clinical protocol. The patients will be recruited from 1.5.2019 to 31.12.2020. The recruited patients will provide both a written informed consent for this study and a Helsinki Biobank consent that covers plasma and surgical samples. Participants can withdraw the consent at any time of the study. The Biobank samples will be taken simultaneously with clinical samples, minimizing the additional harm to participants. A Helsinki University Hospital (HUS) institution review board permission (HUS 60/2019) and ethical statement has been granted (455/2019). The study will be conducted in accordance with the Declaration of Helsinki.

Patients

The patients are recruited prior to surgery from preoperative multidisciplinary team (MDT) meeting. The inclusion criteria into this study is histologically confirmed NSCLC eligible for surgical treatment and naïve for systemic oncological treatments with either formalin-fixed paraffin-embedded tissue or fresh frozen tissue sample available.

The clinical patient data will be collected from electronic medical records (EMR) at each point of time (e.g. preoperative, operative, follow-up). Each patient is evaluated in MDT meetings before and after the surgery, where the both the clinical and the pathological stage is determined. In addition, radiological consolidation/tumor ratio will be calculated from preoperative computerized tomography (CT) scans. This data will be transferred to a secure, certified electronic database (Granitics Unify Med) with access only by group researchers.

Blood and tissue sample collection

The blood and tissue samples will be taken simultaneously with clinical samples. The investigators aim to collect surgically removed tissue samples as well as preoperative and follow-up cfDNA samples from all patients. In addition to surgical samples, tissue samples will be collected from metastatic lesions including autopsy samples in deceased patients. If not already taken, the standard Biobank blood sample will be taken simultaneously to preoperative samples.

Plasma samples will be taken at the time of the patient's clinical blood samples. A preoperative sample will be taken 1-2 day before the surgery. The first post-operative follow-up sample will be taken at the surgical visit 4-6 weeks after the operation. The second and third follow-up samples will be taken at 6 and 12 months during clinical follow-up visit. At each time point, cfDNA samples will be collected into duplicate specialized collection tubes containing fixatives to stabilize DNA from fragmentation (2 x 10ml Streck cfDNA BCT). Blood sample will be centrifuged to extract plasma. Plasma and tissue samples will be stored at -80 celsius in Helsinki Biobank.

Study outcomes Preoperative ctDNA mutations will be matched to clinically important endpoints such as disease-free survival, tumor size, histology, TNM-stage, and overall survival. The clinical cancer recurrence will be obtained from radiological or tumor tissue samples. Disease free survival will be assessed from surgery to disease recurrence in MDT meetings or death. Overall survival is assessed from surgery to death as a result of any cause.

Genetic analysis

Quantitative and mutation specific ctDNA analysis will be made via tumor/somatic exome genome panel that includes 23.000 gene panel with 50 million bases. Germline DNA isolation will be done from buffy coat taken from patients' blood sample (B-Bio-0). Firstly, to achieve true somatic mutations the germline variation is deleted from the ctDNA. Secondly, ctDNA will be compared to tumor tissue DNA mutations to exclude false positive findings. Thirdly, similar or new mutations collected from follow-up samples will be used to detect postsurgical residual disease or cancer recurrence.

The sequencing will be done in collaboration with Institute for Molecular Medicine Finland (FIMM), with their proprietary gene paneling.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria into this study is histologically confirmed NSCLC eligible for surgical treatment and naïve for systemic oncological treatments with either formalin-fixed paraffin-embedded tissue or fresh frozen tissue sample available.

Exclusion Criteria:

* prior metastatic solid cancer, hematological malignancy, known hereditary cancer syndrome, and pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Surgically treated NSCLC patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 2 years
  Lead time to tumor recurrence detection by blood circulating tumor DNA versus clinical recurrence

SECONDARY OUTCOMES:
The concordance of ctDNA and tumor DNA | 1year
  The concordance of mutations detected preoperatively in blood comparing to tumor
Prognostic impact of ctDNA | 4 years
  The correlation of preoperatively or postoperatively collected ctDNA in survival
ctDNA locoregional versus distant recurrence | 4 years
  The difference between locoregional and distant metastasis and findings in postoperative ctDNA
The correlation of ctDNA and clinical features | 2 year
  The correlation of preoperative ctDNA and clinical features such as TNM stage, ECOG class, histopathological features,

CONTACTS AND LOCATIONS:
Overall Officials: Ilkka Ilonen, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: Undecided